CLINICAL TRIAL: NCT00056589
Title: A Phase 1 Escalating Dose Study of the Safety and Pharmacokinetics of Recombinant Factor XIII in Patients With Congenital Factor XIII Deficiency
Brief Title: Safety and Pharmacokinetics of Recombinant Factor XIII in Patients With Congenital Factor Xlll Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F13-1663
Record Dates: First submitted 2003-03-18; First posted 2003-03-20 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Congenital FXIII Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rFXIII (Experimental)
  Interventions: Drug: catridecacog

INTERVENTIONS:
Drug: catridecacog — Single doses of rFXIII administered intravenously (IV) to two subjects in each of the five dose levels (2, 6, 20, 50 and 75 U/kg).

SUMMARY:
This trial was conducted in the United States of America (USA). The aim of this trial was to investigate safety and pharmacokinetics of escalating single doses of catridecacog (recombinant factor XIII, rFXIII) in patients with congenital factor XIII deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Documental congenital FXIII deficiency
* Normal platelet count and clotting parameters
* Adequate renal and hepatic function
* If female and of child-bearing potential, negative serum pregnancy test within 7 days of enrollment
* If a sexually active male or a sexually active female of child-bearing potential, agreement to use a medically accepted form of contraception from the time of enrollment to completion of all follow-up study visits
* Negative drug and alcohol screens

Exclusion Criteria:

* Received blood products or FXIII concentrates within 4 weeks of study enrollment
* Known antibodies to FXIII
* Hereditary or acquired coagulation disorder other than FXIII deficiency
* Previous history of autoimmune disorders involving autoantibodies e.g., systemic lupus erythematosus
* Previous history of thromboembolic events e.g., cerebrovascular accident or deep vein thrombosis or administration of any antithrombotic or antiplatelet drugs within 7 days of study enrollment
* Received treatment with any experimental agent within 30 days of study enrollment
* Any surgical procedure in the 30 days prior to enrollment
* Donated blood within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2003-03; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Days 0-28

SECONDARY OUTCOMES:
Incidence of clinically significant changes from baseline in physical examination or laboratory measurements | Days 0-28
Incidence of rFXIII antibodies, as measured by ELISA (Enzyme-Linked Immuno Sorbent Assay) | Days 0-28
Incidence of yeast antibodies | Days 0-28
FXIII activity measured by the Berichrom® assay | Days 0-28

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Los Angeles, California, United States

REFERENCES:
- [Result] Lovejoy AE, Reynolds TC, Visich JE, Butine MD, Young G, Belvedere MA, Blain RC, Pederson SM, Ishak LM, Nugent DJ. Safety and pharmacokinetics of recombinant factor XIII-A2 administration in patients with congenital factor XIII deficiency. Blood. 2006 Jul 1;108(1):57-62. doi: 10.1182/blood-2005-02-0788. Epub 2006 Mar 23. PMID 16556896
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com